CLINICAL TRIAL: NCT01673698
Title: A Prospective, Randomized Multicenter Study to Evaluate the Safety and Efficacy of the ReShape Duo™ Intragastric Balloon System in Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ReShape Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: The REDUCE Pivotal Trial
Record Dates: First submitted 2012-08-15; First posted 2012-08-28 (Estimated); Results first posted 2015-12-07 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-11

CONDITIONS: Obesity
Keywords: obesity; weight loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ReShape Duo Balloon (Active Comparator): ReShape Duo Balloon
  Interventions: Device: ReShape Duo balloon; Other: Diet counseling; Other: Exercise counseling
- Sham Comparator (Sham Comparator): Sham Comparator
  Interventions: Other: Diet counseling; Other: Exercise counseling

INTERVENTIONS:
Device: ReShape Duo balloon
  Arms: ReShape Duo Balloon
Other: Diet counseling
Other: Exercise counseling

SUMMARY:
The REDUCE Pivotal Trial is a pivotal clinical study designed to develop valid scientific evidence regarding the safety and effectiveness of the ReShape Duo® as an adjunct to diet and exercise in the treatment of obese subjects with one or more obesity-related comorbid conditions.

ELIGIBILITY:
Inclusion criteria:

* Patients 21 to 60 years of age
* Body Mass Index (BMI) ≥ 30 kg/m^2 and ≤ 40 kg/m^2
* At least 5 years of obesity (with BMI ≥ 30)
* Stable weight, defined as a subject who has not gained or lost ≥ 5% of body weight in the 3 months preceding the screening assessment
* Failure to lose weight, within the 36 months preceding the screening date, after participation in either of the following:

  1. A medically or commercially supervised weight loss program involving regular counseling regarding both diet and exercise.
  2. Use of a United States Food and Drug Administration (FDA)-approved diet drug
* The presence of one or more obesity-related comorbid conditions
* Willing and able to provide Informed Consent
* Willing and able to comply with study procedures and visit schedules as specified by the protocol
* If female, the patient must

  1. be postmenopausal for at least 1 year OR
  2. be surgically sterile, OR
  3. if of child bearing potential, must be practicing birth control, be willing to avoid pregnancy for the year of study participation, have a negative serum pregnancy test at screening, and a negative urine pregnancy test at baseline
* Residing within a reasonable distance from the Investigator's treating office and able and willing to travel to the Investigator's office to complete all routine follow-up visits.

Exclusion criteria:

* History of and/or ongoing clinically significant conditions or disorders of the gastrointestinal (GI) tract
* Clinically significant and uncontrolled/unstable hepatic, reproductive, gastrointestinal, renal, hematologic, pulmonary, neurologic, psychiatric, respiratory, endocrine, or cardiovascular system diseases
* Significant acute and/or chronic infections of any kind.
* Severe coagulopathy, hepatic insufficiency or cirrhosis
* Uncontrolled or severe asthma, or any asthma requiring or likely to require inhaled steroid therapy during the anticipated duration of trial participation
* Severe obstructive sleep apnea
* Incompletely controlled hypothyroidism or hyperthyroidism
* Severe systemic disease [consistent with an ASA (American Society of Anesthesia) Physical Status Classification Score of 3 or greater]
* Eating disorders, especially binge eating
* Inability to walk 200 yards without assistance
* Known allergies to any of the device materials or accessories, i.e. silicone, methylene blue, corn starch
* Active drug or alcohol addiction within 12 months of enrollment
* Insulin-dependent diabetes (either Type 1 or Type 2) or a significant likelihood of requiring insulin treatment in the following 12 months
* Depressive disorder with total Beck Depression Inventory (BDI) score > 16 points, and/or BDI affective subscale score > 7 points at screening
* Ongoing treatment, or anticipated need for such treatment, with anticoagulants, known gastric irritants such as aspirin (ASA) or non-steroidal anti-inflammatory drugs (NSAIDs) or agents that can promote gastrointestinal bleeding, within 1 month prior to enrollment, or unwillingness to forego these medications during the study period
* Participation within 60 days of screening date in previous or ongoing clinical trial or current usage of an investigational drug or device
* Any use of an intragastric device prior to this study.
* Genetically caused obesity, such as Prader-Willi syndrome
* Any prior bariatric surgery or likely to undergo bariatric surgery during study follow-up period
* Concomitant use of, or unwillingness to avoid any use of, weight loss medications, weight loss supplements, weight loss herbal preparations and/or participation in any non-study-related organized weight loss program (commercial or medical) at any time during the study, including online or smart phone applications to track or modify food intake, exercise regimens or weight
* Chronic opiate use (> 3 months continuous use) or likely need for opiate use during study participation
* Contraindication or allergy to, or unwillingness to use, proton pump inhibitor medication throughout study follow-up duration-Pregnancy, breast feeding, or intention of becoming pregnant during the study
* Any screening laboratory values outside of the normal range deemed clinically significant by the Investigator
* Anemia defined as either:

  1. Hemoglobin (Hgb) value for females of < 11.0 g/dl, for males < 12.0 g/dl
  2. Abnormal red cell indices and iron deficiency
* Smoking cessation within 3 months of study entry or plans to quit smoking during the study
* Major surgery, open biopsy or significant traumatic injury within 3 months prior to enrollment.
* History of significant adverse experience with sedation or anesthesia
* Serious or uncontrolled psychiatric illness or disorder that could compromise patient understanding of or compliance with study procedures
* Any condition that, in the opinion of the Investigator, would compromise the well-being of the patient or the study or prevent the patient from meeting or performing study requirements, including:

  1. Inability or unwillingness to sign the patient informed consent document.
  2. Inability to participate in all necessary study activities due to physical or mental limitations.
  3. Inability or unwillingness to return for all required follow-up visits.
* Employees/family members of ReShape Medical® or any of its affiliates or contractors
* Employees/family members of the Investigator, sub-Investigators, or their medical office or practice, or surgical, bariatric or hospital organizations at which study procedures may be performed
* An immediate family member (by marriage or blood relationship) of another subject already enrolled in the REDUCE Pivotal Trial

Endoscopic exclusion criteria:

* Peptic ulcerations
* Clinically significant hiatal hernia (> 3 cm)
* Patulous pyloric channel
* Erosive esophagitis
* Varices
* Angiectasias
* Barrett's esophagus
* Esophageal stricture
* Gastric mass
* Any other subject characteristic that would prevent the successful insertion of a ReShape Duo™ or that in the opinion of the Investigator preclude safe use of the ReShape Duo™

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 326 (Actual)
Dates: Start 2012-08; Primary Completion 2014-04 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Lehmann, MD, MPH, Study Director — Lehmann Consulting; Jaime Ponce, MD, Principal Investigator — Hamilton Medical Center
Locations (8):
- United States (8):
  - Scottsdale Healthcare, Scottsdale, Arizona
  - Hamilton Medical Center, Dalton, Georgia
  - Marquette General Surgical Weight Loss Center, Marquette, Michigan
  - University of Minnesota/Department of Gastrointestinal Surgery, Minneapolis, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Greenville Hospital System, Simpsonville, South Carolina
  - Midsouth Bariatrics, Memphis, Tennessee
  - University of TX Health Science Center at Houston, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- ReShape Duo Balloon: ReShape Duo Balloon
  ReShape Duo balloon
  Diet counseling
  Exercise counseling
- Sham Comparator: Sham Comparator
  Diet counseling
  Exercise counseling
Period: Overall Study
Arm/Group | ReShape Duo Balloon | Sham Comparator
Started | 187 | 139
Completed | 136 | 126
Not Completed | 51 | 13
Not completed — Lost to Follow-up | 51 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ReShape Duo Balloon | Sham Comparator | Total
Number analyzed (Participants) | 187 | 139 | 326
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.77 (9.51) | 44.04 (10.17) | 43.88 (9.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178 | 132 | 310
  Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 8 | 23
  Not Hispanic or Latino | 172 | 131 | 303
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 16 | 41
  White | 153 | 118 | 271
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 4 | 12
BMI [Mean (Standard Deviation); unit: kg/m^2] | 35.32 (2.84) | 35.43 (2.63) | 35.37 (2.75)

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Treatment % Excess Weight Loss (EWL) With Control %EWL at Week 24
Description: An inferential test of whether the difference in the mean %EWL between the Treatment and Control groups at 24 weeks was significantly greater than a superiority margin 7.5%.
Time Frame: Week 24
Measure: Mean (Standard Error); unit: percentage of EWL
Groups:
- Treatment: Treatment group
- Control: Control group
Arm/Group | Treatment | Control
Number analyzed (Participants) | 187 | 139
percentage of EWL | 25.1 (1.596) | 11.3 (1.881)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.0041, t-test, 1 sided

2. Primary Outcome: Treatment Group Responder Rate Dichotomized at 25% EWL
Description: An inferential test of whether the percentage of participants in the Treatment Group with a weight loss of >25% EWL at 24 weeks was significantly greater than 35%.
Time Frame: 24 weeks
Population: By design, this trial only studied the weight loss responder rate of the Treatment Group subjects during the first 24 weeks of the study.
Measure: Number; unit: percentage of participants
Groups:
- Intent-to-Treat: Intent-to-Treat population
Arm/Group | Intent-to-Treat
Number analyzed (Participants) | 187
percentage of participants | 48.8
Statistical Analysis 1: Comparison: Intent-to-Treat; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided

3. Secondary Outcome: Weight Loss Maintenance Six Months Following Device Removal
Description: Assess whether significantly greater than 50% of treatment subjects maintained 40% of their excess weight loss at 48 weeks.
Time Frame: 48 weeks
Population: By design, this trial only studied weight loss maintenance at 48 weeks of the Treatment Group who initially received a balloon during the first 24 weeks of the study.
Measure: Number; unit: percentage of participant
Arm/Group | Intent-to-Treat
Number analyzed (Participants) | 156
percentage of participant | 49.4
Statistical Analysis 1: Comparison: Intent-to-Treat; Test type: Superiority or Other; p = 0.5610, Chi-squared

ADVERSE EVENTS:
Time Frame: 24 Weeks
Groups:
- Treatment Subjects: Subjects who were randomized and received a balloon during weeks 0-24
- Control Subjects: Subjects who were randomized to diet and exercise counseling only during weeks 0-24
Arm/Group | Treatment Subjects | Control Subjects
Serious Adverse Events (participants affected / at risk) | 25/187 | 6/139
Other Adverse Events (participants affected / at risk) | 186/187 | 87/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Subjects (N=187) | Control Subjects (N=139)
Vomiting (Gastrointestinal disorders) | 11 (11) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 8 (8) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophageal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pelvic pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal hemmorhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Nervous system disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Subjects (N=187) | Control Subjects (N=139)
Vomiting (Gastrointestinal disorders) | 165 (196) | 7 (7)
Abdominal pain (Gastrointestinal disorders) | 104 (134) | 28 (31)
Nausea (Gastrointestinal disorders) | 110 (124) | 28 (33)
Gastric ulcer (Gastrointestinal disorders) | 72 (73) | 0 (0)
Eructation (Gastrointestinal disorders) | 31 (34) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 28 (32) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 26 (29) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 24 (29) | 7 (7)
Constipation (Gastrointestinal disorders) | 26 (27) | 11 (11)
Abdominal distension (Gastrointestinal disorders) | 20 (21) | 6 (6)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 18 (20) | 3 (3)
Gastritis erosive (Gastrointestinal disorders) | 17 (17) | 0 (0)
Influenza (Infections and infestations) | 7 (7) | 7 (7)
Sinusitis (Infections and infestations) | 6 (6) | 7 (7)
Gastroenteritis viral (Infections and infestations) | 5 (5) | 7 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 24 (26) | 5 (5)
Headache (Nervous system disorders) | 10 (10) | 9 (9)

LIMITATIONS AND CAVEATS:
There are no overall limitations and caveats.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After 12 months after the clinical study report is available, the PI may publish clinical study results, subject to confidentiality agreements and sponsor approval. The PI shall provide sponsor a copy of proposed publication at least 60 days prior to submission so that sponsor may have the opportunity to protect its proprietary rights to information, inventions, or products developed under the clinical study. PI agrees to remove confidential information upon sponsor request.